CLINICAL TRIAL: NCT04459572
Title: The Investigation of Soluble Urokinase Plasminogen Activator Receptor (suPAR) as an Early Indicator of Prognosis and Mortality in Children With Sepsis and Septic Shock: A Prospective Study
Brief Title: As an Early Indicator Biomarker of Prognosis and Mortality in Children With Sepsis and Septic Shock: suPAR
Acronym: suPAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Caner Turan, Director, MD, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TGA-2019-20230
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Septic Shock; Sepsis, Severe
Keywords: sepsis; suPAR; septic shock; children; mortality
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sepsis and sepstic shock (Other): The study consists patients and healty-control group. Patients divided into 3 groups based on severity: sepsis, severe sepsis and septic shock
  Interventions: Diagnostic Test: suPAR

INTERVENTIONS:
Diagnostic Test: suPAR — Soluble Urokinase Plasminogen Activator Receptor (suPAR)

SUMMARY:
The sepsis and septic shock remain major causes of child morbidity and mortality, despite the use of modern antibiotics and resuscitation therapies. Recent interest has focused on biomarkers for early diagnosis, and evaluation the outcomes of sepsis; but there is a still lack of early diagnosis and timely intervention for sepsis in the emergency department (ED). The primary aim was to investigate the role of C-Reactive Protein(CRP), Procalcitonin(PCT), soluble-urokinase plasminogen activator receptor(suPAR) and Presepsin in the early stratification of patients with sepsis. The usefulness of pediatric Sequential Organ Failure Assessment (pSOFA) for predicting of the mortality and the rate of PICU admission in children with septik shock were also investigated. This prospective pilot study was conducted at academic pediatric ED between September 2017-June 2018. All children who met sepsis criteria admitted to ED were involved to study. They kept following up after ED management and their blood samples were taken upon admission on day 0, 1, 2, 4 and 7. The definition made as sepsis, severe sepsis and septic shock. At the same period, 100 healthy children chosen as the control group. The patient characteristics, clinical features, diagnosis, co-morbidities, source of infection, laboratory results (CRP, PCT, lactate, suPAR and Presepsin) and treatments were recorded. The pSOFA score was calculated during first hour of admission. Length of stay in ED and hospital was noted. The main outcome measure was in 7 and 30-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* <18 years
* Admitted to emergency department with sepsis

Exclusion Criteria:

* >18 years
* Diagnosed non-sepsis

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
suPAR values in septic chock | 7 days
  The usefulness of soluble urokinase type plasminogen activator receptor (suPAR) for predicting of the mortality and the rate of PICU admission in children with septik shock

SECONDARY OUTCOMES:
Presepsin level | 7 days
C-Reactive Protein(CRP) level | 7 days
Procalcitonin (PCT) level | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University School of Medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No